CLINICAL TRIAL: NCT03093090
Title: Evaluating Predictive Methods & Product Performance in Healthy Adults for Pediatric Patients, A Case Study: Furosemide
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study never officially began
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2000020010
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Medication Absorption
Keywords: furosemide
MeSH Terms: interventions — Water; Milk; Infant Formula; Ensure Plus; Furosemide

STUDY DESIGN:
Intervention Model Description: A four-way randomized crossover PK study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Water First (Active Comparator): 20mg furosemide administered PO with 6 oz of randomly-assigned study liquid
  Interventions: Dietary Supplement: Water; Dietary Supplement: Parmalat™ Whole Milk; Dietary Supplement: Similac Pro-Advance™; Dietary Supplement: Ensure Plus™; Drug: Furosemide 20 MG
- Milk First (Active Comparator): Parmalat™ Whole Milk 20mg furosemide administered PO with 6 oz of randomly-assigned study liquid
  Interventions: Dietary Supplement: Water; Dietary Supplement: Parmalat™ Whole Milk; Dietary Supplement: Similac Pro-Advance™; Dietary Supplement: Ensure Plus™; Drug: Furosemide 20 MG
- Baby formula first (Active Comparator): Similac Pro-Advance™ 20mg furosemide administered PO with 6 oz of randomly-assigned study liquid
  Interventions: Dietary Supplement: Water; Dietary Supplement: Parmalat™ Whole Milk; Dietary Supplement: Similac Pro-Advance™; Dietary Supplement: Ensure Plus™; Drug: Furosemide 20 MG
- Ensure Plus first (Active Comparator): Ensure Plus™ 20mg furosemide administered PO with 6 oz of randomly-assigned study liquid
  Interventions: Dietary Supplement: Water; Dietary Supplement: Parmalat™ Whole Milk; Dietary Supplement: Similac Pro-Advance™; Dietary Supplement: Ensure Plus™; Drug: Furosemide 20 MG

INTERVENTIONS:
Dietary Supplement: Water — 6 oz
Dietary Supplement: Parmalat™ Whole Milk — 6 oz
  Other Names: Milk
Dietary Supplement: Similac Pro-Advance™ — 6 oz
  Other Names: baby formula
Dietary Supplement: Ensure Plus™ — 6 oz
  Other Names: Ensure
Drug: Furosemide 20 MG — Furosemide is a loop diuretic (water pill) that prevents your body from absorbing too much salt.
  Other Names: Lasix

SUMMARY:
Poorly absorbed medications such as furosemide are common and recent experiments suggest that improvement in absorption can occur if these types of medications are consumed with liquids such as milk. The purpose of this study is to evaluate the absorption of furosemide in normal adults when taken with bottled water, milk (Parmalat™ Whole Milk), baby formula (Similac Pro-Advance™), or Ensure Plus™. These results will be used to make models that predict how these liquids will affect drug absorption in children, potentially providing ways to improve medication absorption in children.

DETAILED DESCRIPTION:
Low solubility drugs are common in the pharmacopeia and it has been estimated that more than 40% of new chemical entities developed by the pharmaceutical industry are practically insoluble in water. Exploratory in vitro studies by the CDER have recently demonstrated that the solubility, and thus potentially the bioavailability, of poorly soluble drugs may be highly enhanced when administered with milk (Parmalat™ Whole Milk) or baby formula (Similac Pro-Advance™).

While the reasons for variable bioavailability of furosemide are not well characterized, the effect of gastric pH, food and dosing liquids are commonly observed on the absorption of BCS Class IV drugs. Absorption variability is much greater in children due to developmental changes in factors such as gastric fluid, blood flow to the intestine, bile acid composition/secretion, intestinal surface area and drug metabolizing enzyme and transporter abundance. Therefore, it is critical to determine the physio-chemical physiological interactions for furosemide that can explain inter-subject and inter-dosing variability. An integrated in vitro, in silico and in vivo pharmacology approach to study the effect of dosing liquids on PK and PD of furosemide is novel. Quantitative understanding of factors affecting furosemide absorption will first be evaluated using in vitro tests such as solubility, dissolution and protein binding with the dosing liquids. The physiochemical information relevant to drug absorption and elimination will be curated from the literature to build the PBPK model. Such in vitro- in vivo extrapolation (IVIVE) linked PBPK modeling approach is crucial to better characterize furosemide's variable bioavailability. Another novel aspect of this study is that we will include renal metabolism of furosemide in the PBPK modeling. While plasma concentration will be critical in determining rate and extent of furosemide absorption, the renal elimination is the primary contributor to the PD response of furosemide as delivery of drug to the luminal surface of the renal tubule is required. PBPK modeling allows extrapolation of model to special population. For example, once the model is optimized and validated to predict effect of dosing liquids on adult PK of furosemide from in vitro data, this approach can be further extrapolated to children using pediatric gut physiological parameters. This novel approach will allow prediction of furosemide PK and PD in children without conducting a clinical study in this difficult to study population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* 4 females and 4 males will be recruited
* Free from known significant chronic medical illness (i.e., hypertension, diabetes, atherosclerosis, chronic kidney disease, liver disease, lupus, taking medications with known interactions with furosemide, a history of syncope/falls, or any acute illness, such as influenza, gastroenteritis, dehydration, electrolyte imbalance, or thrombosis risks).
* Systolic Blood Pressure ≥90 mmHg at Screening Visit

Exclusion Criteria:

* Inability to read English or give informed consent
* Recent hospitalization within 6 months
* Pregnant or lactating
* Allergy or intolerance to furosemide
* Allergy or intolerance to milk, milk products or soy
* Inability to return for 4 consecutive weekly overnight visits at the study site
* Female subjects with low, or borderline low blood pressure, will be evaluated carefully prior to enrollment, to ensure the safety of all subjects involved in the research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
area under the plasma concentration curve | 4 weeks
  The primary analysis will test for overall differences in bioavailability (area under the plasma concentration curve) of furosemide between different liquids. This will be accomplished using a repeated measures ANOVA, or if the distribution is not normally distributed a Wilcoxon-matched pairs sign-rank test.

SECONDARY OUTCOMES:
differences in the peak plasma concentration in furosemide (C-max) | 4 weeks
  Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose. It is a standard measurement in pharmacokinetics. Cmax is the opposite of Cmin, which is the minimum (or trough) concentration that a drug achieves after dosing.
total urinary sodium output | 4 weeks
  collected via urine this is a standard metric of diuretic response

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No